CLINICAL TRIAL: NCT06592365
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Effects and Safety of Green Tea Extract(GTE) Consumption on Blood Glucose Regulation
Brief Title: Clinical Study to Evaluate the Effects and Safety of Green Tea Extract on Blood Glucose Regulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amorepacific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AP-R-2019-01
Record Dates: First submitted 2024-08-20; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Blood Sugar

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GTE (Green tea extract) (Active Comparator): three tablets once daily
  Interventions: Dietary Supplement: GTE
- Placebo (Placebo Comparator): three tablets once daily
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: GTE — oral administration of GTE tablets once daily for 12 weeks
  Arms: GTE (Green tea extract)
Dietary Supplement: Placebo — oral administration of placebo tablets once daily for 12 weeks
  Arms: Placebo

SUMMARY:
This study was conducted to investigate the effects of green tea extracts on reducing blood glucose level

DETAILED DESCRIPTION:
This study was conducted over 12 weeks with a randomized, double-blind, placebo-controlled, parellel design

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged between 19 to 64 years
* BMI between 18.5 and 29.9kg/m²
* fasting blood glucose between 100 and 139 mg/dL (Note: if some subjects with blood glucose range of 126 - 139 mg/dL, those who are taking or requre medication must be excluded to meet ethical standards.)
* subjects who voluntarily decide to participate in this study and sign the informed consent form.

Exclusion Criteria:

* Individuals taking to obesity, dyslipidemia, or uncontrolled hypertension at the screening
* Individuals diagnosed with diabetes and who have taken medications related to blood glucose
* Individuals congenital enzyme deficiencies related to sugar metabolism.
* with hypersensitivity to the test food or ingredients(e.g., green tea, caffeine).
* Individuals ongoing treatment diseases significantly related glucose metabolism.
* Individuals with a history of surgery significantly related to glucose metabolism within the last 6 months
* diagnosed with gastrointestinal diseases, cardiovascular diseases, uncontrolled chronic medical conditions, thyroid disorders, or active malignant tumors requiring medication
* Individuals with liver function impairment or acute or chronic hepatitis or liver cirrhosis
* Individuals with renal disorder
* Individuals with a weight change of 5 kg or more within the last 3 months.

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-08-08 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in fasting glucose level | Baseline, week 12
  blood glucose level detection

SECONDARY OUTCOMES:
changes of indicator of lipid metabolism | Baseline, week 12
  Total cholesterol, HDL, LDL, TG
OGTT | Baseline, week 12
  oral glucose tolerance test
blood biomarkers | Baseline, week 12
  insulin etc.
change in waist circumference(cm) | Baseline, week 12
  -waist circumference was measured using WHO guideline

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Heon Kang, MD, PhD, Principal Investigator — Kangbuk Samsung Hospital
Locations (3):
- South Korea (3):
  - Kangbuk samsung hospital, Seoul
  - Seoul National Universtiy Hospital, Seoul
  - The Catholic University of Korea St. Vincent's Hospital, Seoul